CLINICAL TRIAL: NCT00764335
Title: Unilateral vs Bilateral Total Hip Arthroplasty - the Influence of Medial Femoral Head Offset and Effects on Strength and Aerobic Endurance Capacity
Brief Title: Unilateral vs Bilateral Total Hip Arthroplasty
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: OrtoMedic A/S, Oslo (Unknown); Scandinavian Customized Prosthesis (SCP) (Industry)
Responsible Party: Sponsor
Other Study IDs: 4.2005.1527b
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- unilateral normal: total hip arthroplasty one side, normal offset of medial femoral head
  Interventions: Procedure: total hip arthroplasty one side
- bilateral normal: total hip arthroplasty both sides, normal offset of medial femoral head
  Interventions: Procedure: total hip arthroplasty both sides
- bilateral abnormal offset: total hip arthroplasty both sides, abnormal offset of medial femoral head
  Interventions: Procedure: total hip arthroplasty both sides
- controls: Healthy, age-matched control group

INTERVENTIONS:
Procedure: total hip arthroplasty one side — unilateral total hip arthroplasty
  Groups: unilateral normal
Procedure: total hip arthroplasty both sides — bilateral total hip arthroplasty
  Groups: bilateral abnormal offset; bilateral normal

SUMMARY:
The purpose of the present study was to determine whether unilaterally operated total hip arthroplasty (THA) patients were superior to bilaterally operated THA patients with respect to aerobic endurance capacity, muscle strength and gait patterns 3-5 years after surgery, and to what extent medial femoral head offset (FO) influenced hip abductor strength.

ELIGIBILITY:
Inclusion Criteria:

* Undergone hip surgery 3-5 years ago
* Age < 70 years

Exclusion Criteria:

* Heart or lung diseases
* Malign diseases
* No muscle/skeletal diseases that compromises testing

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects selected from orthopaedic out-patient department
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Hoff, PhD prof, Study Director — Norwegian University of Science and Technology

REFERENCES:
- [Result] Husby VS, Bjorgen S, Hoff J, Helgerud J, Benum P, Husby OS. Unilateral vs. bilateral total hip arthroplasty - the influence of medial femoral head offset and effects on strength and aerobic endurance capacity. Hip Int. 2010 Apr-Jun;20(2):204-14. doi: 10.1177/112070001002000211. PMID 20544648